CLINICAL TRIAL: NCT05169606
Title: Effect of Tissue Flossing, Active Isolated Stretch, Proprioceptive Neuromuscular Facilitation on Hamstring Among Knee Osteoarthritis Patients
Brief Title: Effect of Tissue Flossing, AIS, PNF on Hamstring Among Knee OA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01068 Mohammad Jawwad
Record Dates: First submitted 2021-12-13; First posted 2021-12-27 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis
Keywords: Tissue Flossing; Active Isolated Stretch; Proprioceptive Neuromuscular Facilitation; Knee Osteoarthritis; Pain; Range of motion
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tissue Flossing (Experimental): Tissue flossing is a technique that requires wrapping of a thick rubber band around a joint or muscle concomitantly performing ROM tasks for 1-3 minutes. The results include increase in range of motion and a decrease in pain of the effected muscles. The phenomenon behind getting results through this technique is hypothesized to be blood reperfusion to an occluded area via tissue flossing augments exercise performance mechanisms such as growth hormone, catecholamine responses, muscle force contractility and the efficiency of excitation-contraction coupling in the muscles. In addition, tissue flossing may influence fascia tightness via the fascial mechanoreceptors, therefore reducing muscle activity, resulting in a greater ROM. Nevertheless, the underlying mechanism for tissue flossing, these mechanisms remain speculative.
  Interventions: Other: Tissue Flossing; Other: Active Isolated Stretch; Other: Proprioceptive Neuromuscular Facilitation
- Active Isolated Stretch (Experimental): Active Isolated Stretch is a specific stretching program developed by Aaron Mattes over 30 years ago. Active isolated stretch is also found to be effective to increase flexibility and improve ROM.
  Interventions: Other: Tissue Flossing; Other: Active Isolated Stretch; Other: Proprioceptive Neuromuscular Facilitation
- Proprioceptive Neuromuscular Facilitation (Experimental): Proprioceptive neuromuscular facilitation (PNF) technique has already been found to have beneficial effects in improving hamstring flexibility and reducing pain in the knee joint of knee OA patients.
  Interventions: Other: Tissue Flossing; Other: Active Isolated Stretch; Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: Tissue Flossing — Tissue flossing is a technique that requires wrapping of a thick rubber band around a joint or muscle concomitantly performing ROM tasks for 1-3 minutes. The results include increase in range of motion and a decrease in pain of the effected muscles. The phenomenon behind getting results through this technique is hypothesized to be blood reperfusion to an occluded area via tissue flossing augments exercise performance mechanisms such as growth hormone, catecholamine responses, muscle force contractility and the efficiency of excitation-contraction coupling in the muscles. In addition, tissue flossing may influence fascia tightness via the fascial mechanoreceptors, therefore reducing muscle activity, resulting in a greater ROM. Nevertheless, the underlying mechanism for tissue flossing, these mechanisms remain speculative.
Other: Active Isolated Stretch — AIS is a specific stretching program developed by Aaron Mattes. This technique is based on these four basic principles:
  Isolate the muscle to be stretched. Repeat the stretch eight to 10 times. Hold each stretch for no more than two seconds. Exhale on the stretch; inhale on the release.
Other: Proprioceptive Neuromuscular Facilitation — Proprioceptive neuromuscular facilitation (PNF) technique has already been found to have beneficial effects in improving hamstring flexibility and reducing pain in the knee joint of knee OA patients

SUMMARY:
Tissue flossing has been known to produce results such as pain relief and improved range of motion, this technique might yield positive results in knee OA patients as well. These effects can further be compared with existing treatment method for treatment of hamstring such as Active isolated stretch and Proprioceptive Neuromuscular facilitation. This study will be among the first to carry out the technique of flossing in knee OA patients.

DETAILED DESCRIPTION:
Arthritis is a broad term that encompasses a large number of diseases that affects one or more joints of the body. Amongst all other forms, Osteoarthritis (OA) is the most prevalent. Osteoarthritis is widespread throughout the world. It is one of the top leading causes of disability on a global scale. Previously this disease was thought to simply be due to biomechanical disturbances causing 'wear and tear' thus giving the characteristic feature of articular destruction leading to stiffness, inflammation and loss of mobility of joints over a long period of time. Due to recent advances in this area of study, evidence has revealed that OA has a collection of a much more complex multifactorial process composed of inflammatory and metabolic factors.

Typical clinical symptoms found in patients with Osteoarthritis include severe joint pain, stiffness, and significantly reduced mobility, which leads to decreased productivity and quality of life among the patients . Osteoarthritis can develop in any joint of the human body but the most frequently affected are the knees, hips, hands, facet joints and feet. This disease not only has an impact on the patient but in addition it also gives rise to an increased socioeconomic burden on the society. In 2005, it was estimated that over 26 million people in the USA had some form of OA. An estimated 30.8 million adults in the United States and 300 million individuals worldwide are living with OA. The severity of the Osteoarthritis can be categorized according Kellgren-Lawrence Grading System for Osteoarthritis.

Osteoarthritis frequently affects the weight bearing joints of the body. Knee OA has a high prevalence and is a disabling joint disease. The OA of the knee joint almost accounts for more than 80% of the disease's total burden and it affects no less than 19% of American adults aged 45 years and older. The knee joint Osteoarthritis is not only more important for its high prevalence rate in comparison to other types of OA but also for its presentation at earlier age groups. The incidence of knee OA increases by age and further increases with longer lifetime. The prevalence is found to be higher in females as compared to males. Participation in sports, injury to the joint, high BMI, and genetic susceptibility are also some factors that predispose individuals to the development of Knee osteoarthritis. Previous knee trauma increases the risk of knee OA 3.86 times. Overall an estimate of 80% of patients with knee OA suffer from some form of movement restriction, while 20% are unable to perform basic daily activities; indeed, 11% of sufferers require personal care. Amongst the cardinal symptoms of OA, pain is the biggest concern, and motor disability and impaired proprioception are important secondary factors.

Proprioceptive neuromuscular facilitation (PNF) technique has already been found to have beneficial effects in improving hamstring flexibility and reducing pain in the knee joint of knee OA patients. Active isolated stretch is also found to be effective to increase flexibility and improve ROM.

Tissue flossing is a relatively new technique to be introduced in the world of research. Tissue flossing is a new method that aims to improve range of motion (ROM), reduce pain, prevent injury, or enhance recovery. Since its arrival the technique has been researched upon mainly on the athletic population. Tissue flossing is a technique that requires wrapping of a thick rubber band around a joint or muscle concomitantly performing ROM tasks for 1-3 minutes. The results include increase in range of motion and a decrease in pain of the effected muscles. The phenomenon behind getting results through this technique is hypothesized to be blood reperfusion to an occluded area via tissue flossing augments exercise performance mechanisms such as growth hormone, catecholamine responses, muscle force contractility and the efficiency of excitation-contraction coupling in the muscles. In addition, tissue flossing may influence fascia tightness via the fascial mechanoreceptors, therefore reducing muscle activity, resulting in a greater ROM. Nevertheless, the underlying mechanism for tissue flossing, these mechanisms remain speculative.

ELIGIBILITY:
Inclusion Criteria:

* Grade 1 and Grade 2 osteoarthritis patients
* Tight Hamstrings (pain in passive Straight Leg Raise <70 degrees)
* Willing to participate

Exclusion Criteria:

* Patients who have latex allergy
* Hypertension (i.e., resting systolic 130-159 mm Hg and diastolic 85-99 mm Hg)
* Venous thrombotic disease
* Heart diseases
* Respiratory diseases apparent neurological, dermatitis, or neurological problems in their legs
* Patients who do not give consent.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Straight Leg Raise for Flexibility | for four weeks
  The leg is raised straight raise test when performed when the subject is placed supine, the therapist grasps the ankle and lifts the leg straight up, while stabilises the same anterior superior iliac spine. If the leg cannot be raised beyond 80degrees the hamstrings is considered tight.
Passive Knee Extension Test for Flexibility | For four weeks
  The patient is positioned in supine with the hip of the tested leg in 90 degrees of flexion.The contralateral leg stays flat on the examination table. The clinician extends the knee until reaching the maximal tolerable stretch of the hamstring muscle as indicated by the patient with the ipsilateral hip remaining in 90 of flexion. The knee angle is then measured with a goniometer.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | For four weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The test-retest reliability of the WOMAC varies for the different subscales.
Numeric pain rating scale for pain | for four weeks
  Numeric pain rating scale is used to capture the patient's level of pain. Patients will be asked to indicate the intensity of current, best, and worst levels of pain over the past 24 hours using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Alees Medical centre, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No